CLINICAL TRIAL: NCT02090452
Title: Telemedical Solutions in Medical Emergencies, Advantages and Disadvantages for Patients, Healthcare Professionals, and the Healthcare System: Study 1: "Mobile Transmission of Prehospital Vital Signs to the Emergency Department - Effect on Patient Outcomes, Treatment and Diagnosis"
Brief Title: Mobile Transmission of Prehospital Vital Signs to the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Central Denmark Region (Other)
Responsible Party: Principal Investigator, Nikolaj Raaber, MD, University of Aarhus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NRAA
Record Dates: First submitted 2014-02-20; First posted 2014-03-18 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Telemedicine; Triage; Emergency Medical Service
Keywords: Telemedicine; Mobile; Vital signs; Prehospital care; Emergency medicine
MeSH Terms: interventions — Vital Signs; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transmission of vital signs, ecg, chat (Experimental): Data from patients transported in ambulances with equipment which enables real time transmission of vital signs, ecg and chat from ambulances to the emergency department.
  Interventions: Device: Real time transmission of patient related data. Device used: MobiMed 3.1, manufactured by Ortivus AB Sweden
- No transmission of data (No Intervention): Patient transported with conventional ambulances without the possibility to transmit real time patient related data.

INTERVENTIONS:
Device: Real time transmission of patient related data. Device used: MobiMed 3.1, manufactured by Ortivus AB Sweden
  Other Names: Vital signs, ECG and Chat-messaging delivered real time from prehospital ambulances to the receiving emergency dept.
  Arms: Transmission of vital signs, ecg, chat

SUMMARY:
The purpose of this study is to examine if real time transmission of vital signs, ECG and chat communication between the prehospital ambulances and the emergency department has an effect on patient mortality, ICU admission, hospitalization time, time to doctor, time to treatment and time to diagnostics

ELIGIBILITY:
Inclusion Criteria:

* All patients transported with ambulance to the emergency department

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time to physician | Time from arrival to first patient-physician contact, assessed up to 36 months
  Time from the patient arrival registered in the patients' logistics system (Cetrea) to registered first patient/physician contact registered in the same patients logistics system.

SECONDARY OUTCOMES:
All cause mortality | 30 days, assessed up to 36 months
Time to treatment | Time from arrival to administration of first iv. antibiotics, assessed up to 36 months
  Time from the patient arrival registered in the patients' logistics system (Cetrea) to first administered iv antibiotics registered in the patient's hospital record
Time to x-ray | Time form arrival at the emergency department to completion of x-ray requisition form, assessed up to 36 months
  Time from the patient arrival registered in the patients' logistics system (Cetrea) to completion of x-ray requisition form registered in the radiologic logistics system (Kodak RIS, 2010 edition)
Time to ICU | Time from arrival to admission to the ICU, assessed up to 36 months
  Time from the patient arrival registered in the patients' logistics system (Cetrea) to time of admission to the ICU registered in the patient's hospital record. .
Number of ICU admissions | During present hospitalization, assessed up to 36 months

OTHER OUTCOMES:
Emergency department staff evaluation of usability of equipment | At the time of using the equipment, assessed up to 36 months
  The staff at the emergency department fill out a survey after the use of the equipment which provides ecg, vital signs, chat.
Ambulance staff evaluation of usability of equipment | At the time of using the equipment, assessed up to 36 months
  The ambulance staff fill out a survey after the use of the equipment which provides ecg, vital signs, chat.

CONTACTS AND LOCATIONS:
Overall Officials: Erika F. Christensen, MD, Medical director, Study Director — Central Denmark Region
Locations (3):
- Denmark (3):
  - Prehospital Emergency Medical Services, Aarhus, Central Denmark Region, Aarhus N
  - Horsens Regional Hospital, Central Region Denmark, Horsens
  - Responce A/S, Horsens